CLINICAL TRIAL: NCT01028963
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of CCX140-B in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety and Efficacy of CCX140-B in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL004_140
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; CCX140-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Active control (Active Comparator)
  Interventions: Drug: pioglitazone
- Active Study Medication (Group C) (Experimental): CCX140-B
  Interventions: Drug: CCX140-B
- Active Study Medication (Group D) (Experimental): CCX140-B
  Interventions: Drug: CCX140-B

INTERVENTIONS:
Drug: Placebo — Placebo capsules once daily
  Arms: Placebo
Drug: pioglitazone — pioglitazone 30 mg tablet once daily
  Arms: Active control
Drug: CCX140-B — CCX140-B capsules once daily (Group C)
  Arms: Active Study Medication (Group C)
Drug: CCX140-B — CCX140-B capsules once daily (Group D)
  Arms: Active Study Medication (Group D)

SUMMARY:
The purpose of this study is to evaluate the safety and potential effectiveness of CCX140-B in subjects with Type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of CCX140-B in subjects with Type 2 diabetes mellitus (T2DM) based on subject incidence of adverse events.

The secondary objectives of this study include evaluation of the effect of CCX140-B on several measures of effectiveness commonly used in the evaluation of diabetes medications.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed type 2 diabetes mellitus
* Must have a body mass index ≥25 and <45 kg/m2, but if body mass index is ≥25 and <28 kg/m2, then waist circumference must be >94 cm for men and >80 cm for women
* Must be on a stable dose of metformin for at least 8 weeks prior to randomization
* Hemoglobin A1c (HbA1c) of 6.5 to 10.0% inclusive and fasting plasma glucose 135 to 270 mg/dL inclusive at Screening

Key Exclusion Criteria:

* Type 1 diabetes mellitus or history of diabetic ketoacidosis
* Received insulin treatment within 12 weeks of randomization
* Received chronic (more than 7 days) systemic glucocorticoid treatment within 12 weeks of randomization
* Received sulfonylurea, thiazolidinedione, exenatide, or any other glucose lowering treatment (other than metformin) within 8 weeks of randomization
* Symptomatic congestive heart failure requiring prescription medication, clinically evident peripheral edema, poorly-controlled hypertension (systolic blood pressure >160 or diastolic blood pressure >100), history of unstable angina, myocardial infarction or stroke within 6 months of randomization, or chronic renal failure
* History or presence of drug-induced myopathy, drug-induced creatine kinase elevation, or leukopenia (WBC count <3.5 x 10(9)/L)
* History or presence of any form of cancer within the 5 years prior to randomization, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis
* Fasting serum triglyceride >400 mg/dL

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events | 28 days

SECONDARY OUTCOMES:
Effect on fasting plasma glucose concentration | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (28):
- Australia (2):
  - Auchenflower, Queensland
  - Kippa-Ring, Queensland
- Czechia (12):
  - Beroun
  - Hlučín
  - Neratovice
  - Nový Jičín
  - Ostrava
  - Pardubice
  - Prague
  - Přelouč
  - Slaný
  - Uherský Brod
  - Uničov
  - Ústí nad Labem
- Germany (8):
  - Basenheim
  - Berlin
  - Cologne
  - Dresden
  - Heidelberg
  - Mannheim
  - Nuremberg
  - Saarlouis
- Hungary (4):
  - Balatonfüred
  - Budapest
  - Sátoraljaújhely
  - Szikszó
- New Zealand (2):
  - Christchurch
  - Wellington